CLINICAL TRIAL: NCT05862337
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Phase 3 Study of Anlotinib Hydrochloride Capsules Combined With Penpulimab Injection in Patients With High Risk of Relapse After Radical Surgery or Ablation of Hepatocellular Carcinoma (HCC).
Brief Title: Anlotinib Hydrochloride Capsules Combined With Penpulimab Injection for the Treatment of Hepatocellular Carcinoma at High Risk of Recurrence.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALTN-AK105-III-06
Record Dates: First submitted 2023-05-15; First posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2022-07

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — penpulimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anlotinib hydrochloride capsules + Penpulimab injection (Experimental): Anlotinib hydrochloride capsules + Penpulimab injection, 21 days as a treatment cycle.
  Interventions: Drug: Anlotinib hydrochloride capsules, Penpulimab injection
- Anlotinib hydrochloride capsules -matching placebo+ Penpulimab injection -matching placebo (Placebo Comparator): Anlotinib hydrochloride capsules -matching placebo+ penpulimab injection -matching placebo, 21 days as a treatment cycle.
  Interventions: Drug: Anlotinib hydrochloride capsules -matching placebo, Penpulimab injection -matching placebo

INTERVENTIONS:
Drug: Anlotinib hydrochloride capsules, Penpulimab injection — Anlotinib hydrochloride capsules is a multitargeted receptor tyrosine kinase inhibitor.
  Penpulimab injection is a humanized monoclonal antibody targeting programmed cell death protein 1 (PD-1).
  Arms: Anlotinib hydrochloride capsules + Penpulimab injection
Drug: Anlotinib hydrochloride capsules -matching placebo, Penpulimab injection -matching placebo — placebo control, no active substance.
  Arms: Anlotinib hydrochloride capsules -matching placebo+ Penpulimab injection -matching placebo

SUMMARY:
The primary objective of this study was to evaluate the efficacy of anlotinib hydrochloride capsules combined with penpulimab injection (test group) versus placebo (control group) for adjuvant therapy after radical surgery or ablation in HCC patients with high risk of recurrence by assessing recurrence-free survival (RFS).

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-75 years old; Eastern Cooperative Oncology Group Performance Status (ECOG PS) ≤ 1; Predicted survival ≥12 weeks.
* Subjects with hepatocellular carcinoma (HCC) confirmed by histopathology or cytology or who meet the diagnostic criteria for Primary Liver Cancer 2022 or the American Association for the Study of Hepatology (AASLD) hepatocellular carcinoma.
* Subjects who received radical excision or ablation (Radio Frequency Ablation (RFA) or Microwave Ablation (MWA) only) within 4 to 12 weeks prior to randomization (multiple modalities or combined or multiple treatments are not acceptable).
* No major vena portae 3 (Vp3) or vena portae 4 (Vp4) in the portal vein or any level of vascular invasion in the hepatic vein or inferior vena cava.
* No extrahepatic metastasis.
* High risk factors for recurrence after radical resection or complete ablation.
* Complete recovery from surgical resection or ablation within 4 weeks before randomization.

Exclusion Criteria:

* Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC histology.
* Evidence of residual, recurrent, or metastatic disease at randomization.
* More than one surgical treatment for hepatocellular carcinoma; Received more than 1 prophylactic Transcatheter Arterial Chemoembolization (TACE) treatment after surgery; or received Hepatic Artery Infusion Chemotherapy (HAIC) therapy after surgery.
* Previous use of antiangiogenic drugs or PD-1, Programmed Cell Death-Ligand 1 (PD-L1) and other related immunotherapy drugs or systemic chemotherapy drugs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival (RFS) | Baseline up to 3 years.
  RFS assessed by the Blinded Independent Image Review Committee and the investigator is the time from randomization to the first local, regional recurrence or distant metastasis, or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
Time to recurrence(TTR) | Baseline up to 3 years.
  TTR assessed by the Blinded Independent Image Review Committee and the investigator is the time from randomization to the first local, regional recurrence or distant metastasis, whichever occurred first.
Time to extrahepatic metastasis or macrovascular invasion | Baseline up to 3 years.
  Time to extrahepatic metastasis or macrovascular invasion as assessed by the investigator.
Overall survival (OS) | Baseline up to 3 years.
  OS defined as the time from the date of randomization until the date of death due to any cause.
Objective response rate (ORR) after first recurrence | Baseline up to 3 years.
  subjects with evaluable tumor lesion status who were cross-treated with Anlotinib hydrochloride capsules combined with Penpulimab injection developed complete response or partial response after a first HCC relapse as assessed by Response Evaluation Criteria In Solid Tumors (RECIST) v1.1.

CONTACTS AND LOCATIONS:
Locations (67):
- China (67):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Anhui Provincial Hospital, Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Beijing Friendship hospital of Capital Medical University, Beijing, Beijing Municipality
  - Beijing YouAn Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Chongqing University Three Gorges Hospital, Chongqing, Chongqing Municipality
  - Mengchao Hepatobiliary Hospital of Fujian Medical, Fuzhou, Fujian
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Gansu Provincial Cancer Hospital, Lanzhou, Gansu
  - Lanzhou University First Hospital, Lanzhou, Gansu
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - Gansu Provincial Hospital, Lanzhou, Gansu
  - Guangdong People's Hospital, Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning, Guangxi
  - Guizhou Provincial People'S Hospital, Guiyang, Guizhou
  - The Affiliated Cancer Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Affiliated Hospital Of Zunyi Medical University, Zunyi, Guizhou
  - Hainan Provincial People's Hospital, Haikou, Hainan
  - The Second Affiliated Hospital of Hainan Medical University, Haikou, Hainan
  - Affiliated Cancer Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - The Third Xiang Ya Hospital of Central South University, Changsha, Hunan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Chifeng Municipal Hospital, Chifeng, Inner Mongolia
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - Jiangsu Province People's Hospital, Nanjing, Jiangsu
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - Nantong Tumor Hospital, Nantong, Jiangsu
  - Ganzhou People's Hospital, Ganzhou, Jiangxi
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - The Second Hospital of Dalian Medical University, Dalian, Liaoning
  - The First Affiliated Hospital of Jinzhou Medical University, Jinzhou, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - The Sixth People's Hospital of Shen Yang, Shenyang, Liaoning
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - Binzhou Medical University Hospital, Binzhou, Shandong
  - Shandong Cancer Hospital, Jinan, Shandong
  - The First Affiliated Hospital of Naval Medical University, Shanghai, Shanghai Municipality
  - Third Affiliated Hospital of Naval Medical University, Shanghai, Shanghai Municipality
  - Baoji Central Hospital, Baoji, Shanxi
  - Heping Hospital Affiliated to Changzhi Medical College, Changzhi, Shanxi
  - The Second Affiliated Hospital of Air Force Medical University, Xi’an, Shanxi
  - First Affiliated Hospital of Xian Jiaotong University, Xi’an, Shanxi
  - Xi'an International Medical Center Hospital, Xi’an, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan
  - Affiliated Hospital Of North Sichuan Medical College, Nanchong, Sichuan
  - Tianjin Third Central Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Tianjin Cancer Hospital Airport Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Sir Run Run Shaw Hospital Zhetiang University School of Medicine, Hangzhou, Zhejiang
  - Ningbo Medical Center Lihuili Hospital, Ningbo, Zhejiang
  - Shaoxing People's Hospital, Shaoxing, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang